CLINICAL TRIAL: NCT05738343
Title: Adesione Alla Dieta Mediterranea Dei Pazienti Pediatrici Affetti Dalla Sindrome Dell'Intestino Irritabile (IBS): Studio Pilota
Brief Title: Dieta Mediterranea e Sindrome Dell'Intestino Irritabile in Pazienti Pediatrici
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Di Nardo, Professor, University of Roma La Sapienza
Other Study IDs: CE 6885/2022
Record Dates: First submitted 2023-01-24; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; pediatric; mediterranean diet; childhood; ibs; treatment
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens | interventions — Diet, Mediterranean

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dieta mediterranea — nutritional education or Mediterranean food scheme
  Other Names: mediterranean diet

SUMMARY:
The goal of this observational study is to observe pediatric patients with IBS (irritable bowel syndrome). The main question it aims to answer are:

* adherence to the Mediterranean diet of children with IBS
* in patients not adhering to the Mediterranean diet, evaluate the efficacy of the nutritional intervention Participants will be visited, blood samples will be taken, abdomen ultrasound and they will answer questionnaires.

DETAILED DESCRIPTION:
The goal of this observational study is to observe pediatric patients with IBS (irritable bowel syndrome). the diagnosis of IBS will be placed in reference to the Rome IV criteria. To make a diagnosis, at least 2 of:

* abdominal pain for at least 4 days per month associated with one or more of: pain associated with bowel movements, change in bowel frequency, change in stool consistency must be present.
* In children with constipation, pain persists as the constipation resolves.
* The symptoms are not explained by another medical condition. Participants will be visited, blood samples will be taken, abdomen ultrasound if necessary will be performed and they will answer questionnaires.

The main question it aims to answer are:

* adherence to the Mediterranean diet of children with IBS
* in patients not adhering to the Mediterranean diet, evaluate the efficacy of the nutritional intervention. if BMI between 5 and 85, nutritional education will be carried out for a healthy and correct diet. If BMI between 85 and 95 or greater than 95, personalized Mediterranean food scheme.

ELIGIBILITY:
Inclusion Criteria:

- diagnosis of IBS, based on Rome IV criteria.

Exclusion Criteria:

* use of NSAIDs in the last 3 months;
* allergies or intolerances;
* recent diagnosis (last 3 months) of bacterial or parasitic infections of the gastrointestinal tract;
* psychiatric diseases;
* chronic inflammatory diseases of the gastrointestinal tract.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients belonging to the Sant'Andrea hospital pediatric gastroenterology clinic, in Rome.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
pediatric patients with IBS adherence to the Mediterranean diet | Day 0
  adherent patients on enrolled patients

SECONDARY OUTCOMES:
How many pediatric IBS patients who do not adhere to the Mediterranean diet, respond to nutritional intervention? | Day 7
  Pediatric IBS patients who do not adhere to the Mediterranean diet will be instructed in a correct diet according to the Mediterranean diet or they will have a personalized diet and then the Rome IV criteria will be re-evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Di Nardo, Principal Investigator — Sapienza, Università di Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devanarayana NM, Rajindrajith S. Irritable bowel syndrome in children: Current knowledge, challenges and opportunities. World J Gastroenterol. 2018 Jun 7;24(21):2211-2235. doi: 10.3748/wjg.v24.i21.2211. PMID 29881232
- [Background] Cassar GE, Youssef J G, Knowles SR, Moulding R, Austin D. The Impact of Diagnostic Status on Quality of Life in Irritable Bowel Syndrome. Turk J Gastroenterol. 2021 Oct;32(10):808-818. doi: 10.5152/tjg.2021.20517. PMID 34787085
- [Background] Hyams JS, Di Lorenzo C, Saps M, Shulman RJ, Staiano A, van Tilburg M. Functional Disorders: Children and Adolescents. Gastroenterology. 2016 Feb 15:S0016-5085(16)00181-5. doi: 10.1053/j.gastro.2016.02.015. Online ahead of print. PMID 27144632
- [Background] Saps M, Miranda A. Gastrointestinal Pharmacology. Handb Exp Pharmacol. 2017;239:147-176. doi: 10.1007/164_2016_119. PMID 28236087
- [Background] Saps M, Biring HS, Pusatcioglu CK, Mintjens S, Rzeznikiewiz D. A comprehensive review of randomized placebo-controlled pharmacological clinical trials in children with functional abdominal pain disorders. J Pediatr Gastroenterol Nutr. 2015 May;60(5):645-53. doi: 10.1097/MPG.0000000000000718. PMID 25906454
- [Background] Bhesania N, Cresci GAM. A nutritional approach for managing irritable bowel syndrome. Curr Opin Pediatr. 2017 Oct;29(5):584-591. doi: 10.1097/MOP.0000000000000536. PMID 28737582
- [Background] Paduano D, Cingolani A, Tanda E, Usai P. Effect of Three Diets (Low-FODMAP, Gluten-free and Balanced) on Irritable Bowel Syndrome Symptoms and Health-Related Quality of Life. Nutrients. 2019 Jul 11;11(7):1566. doi: 10.3390/nu11071566. PMID 31336747
- [Background] Iaccarino Idelson P, Scalfi L, Valerio G. Adherence to the Mediterranean Diet in children and adolescents: A systematic review. Nutr Metab Cardiovasc Dis. 2017 Apr;27(4):283-299. doi: 10.1016/j.numecd.2017.01.002. Epub 2017 Jan 12. PMID 28254269
- [Background] Manzano-Carrasco S, Felipe JL, Sanchez-Sanchez J, Hernandez-Martin A, Gallardo L, Garcia-Unanue J. Weight Status, Adherence to the Mediterranean Diet, and Physical Fitness in Spanish Children and Adolescents: The Active Health Study. Nutrients. 2020 Jun 4;12(6):1680. doi: 10.3390/nu12061680. PMID 32512886
- [Background] Serra-Majem L, Tomaino L, Dernini S, Berry EM, Lairon D, Ngo de la Cruz J, Bach-Faig A, Donini LM, Medina FX, Belahsen R, Piscopo S, Capone R, Aranceta-Bartrina J, La Vecchia C, Trichopoulou A. Updating the Mediterranean Diet Pyramid towards Sustainability: Focus on Environmental Concerns. Int J Environ Res Public Health. 2020 Nov 25;17(23):8758. doi: 10.3390/ijerph17238758. PMID 33255721
- [Background] Mannocci A, Di Thiene D, Del Cimmuto A, Masala D, Boccia A, De Vito E, La Torre G. International Physical Activity Questionnaire: validation and assessment in an Italian sample. Ital J Public Health 2010; 7(4):369-76.
- [Background] Veiga OL, Gomez-Martinez S, Martinez-Gomez D, Villagra A, Calle ME, Marcos A; AFINOS Study Group. Physical activity as a preventive measure against overweight, obesity, infections, allergies and cardiovascular disease risk factors in adolescents: AFINOS Study protocol. BMC Public Health. 2009 Dec 19;9:475. doi: 10.1186/1471-2458-9-475. PMID 20021690
- [Background] Zanini B, Simonetto A, Bertolotti P, Marullo M, Marconi S, Becchetti C, Gilioli G, Valerio A, Donato F, Ricci C, Castellano M. A new self-administered semi-quantitative food frequency questionnaire to estimate nutrient intake among Italian adults: development design and validation process. Nutr Res. 2020 Aug;80:18-27. doi: 10.1016/j.nutres.2020.05.008. Epub 2020 May 19. PMID 32673962
- [Background] Archero F, Ricotti R, Solito A, Carrera D, Civello F, Di Bella R, Bellone S, Prodam F. Adherence to the Mediterranean Diet among School Children and Adolescents Living in Northern Italy and Unhealthy Food Behaviors Associated to Overweight. Nutrients. 2018 Sep 18;10(9):1322. doi: 10.3390/nu10091322. PMID 30231531
- [Background] Bonaccorsi G, Furlan F, Scocuzza M, Lorini C. Adherence to Mediterranean Diet among Students from Primary and Middle School in the Province of Taranto, 2016-2018. Int J Environ Res Public Health. 2020 Jul 28;17(15):5437. doi: 10.3390/ijerph17155437. PMID 32731568
- [Background] Trapanotto M, Giorgino D, Zulian F, Benini F, Varni JW. The Italian version of the PedsQL in children with rheumatic diseases. Clin Exp Rheumatol. 2009 Mar-Apr;27(2):373-80. PMID 19473585
- [Background] Gallagher D, Andres A, Fields DA, Evans WJ, Kuczmarski R, Lowe WL Jr, Lumeng JC, Oken E, Shepherd JA, Sun S, Heymsfield SB. Body Composition Measurements from Birth through 5 Years: Challenges, Gaps, and Existing & Emerging Technologies-A National Institutes of Health workshop. Obes Rev. 2020 Aug;21(8):e13033. doi: 10.1111/obr.13033. Epub 2020 Apr 20. PMID 32314544
- [Background] Van Eyck A, Eerens S, Trouet D, Lauwers E, Wouters K, De Winter BY, van der Lee JH, Van Hoeck K, Ledeganck KJ. Body composition monitoring in children and adolescents: reproducibility and reference values. Eur J Pediatr. 2021 Jun;180(6):1721-1732. doi: 10.1007/s00431-021-03936-0. Epub 2021 Jan 22. PMID 33481106
- [Background] Dos Santos RRG, Forte GC, Mundstock E, Amaral MA, da Silveira CG, Amantea FC, Variani JF, Booij L, Mattiello R. Body composition parameters can better predict body size dissatisfaction than body mass index in children and adolescents. Eat Weight Disord. 2020 Oct;25(5):1197-1203. doi: 10.1007/s40519-019-00750-4. Epub 2019 Jul 23. PMID 31338791
- [Background] Orsso CE, Gonzalez MC, Maisch MJ, Haqq AM, Prado CM. Using bioelectrical impedance analysis in children and adolescents: Pressing issues. Eur J Clin Nutr. 2022 May;76(5):659-665. doi: 10.1038/s41430-021-01018-w. Epub 2021 Oct 7. PMID 34620999
- [Background] Guida B, Pietrobelli A, Trio R, Laccetti R, Falconi C, Perrino NR, Principato S, Pecoraro P. Body mass index and bioelectrical vector distribution in 8-year-old children. Nutr Metab Cardiovasc Dis. 2008 Feb;18(2):133-41. doi: 10.1016/j.numecd.2006.08.008. Epub 2007 Feb 16. PMID 17307345
- [Background] Savino F, Cresi F, Grasso G, Oggero R, Silvestro L. The Biagram vector: a graphical relation between reactance and phase angle measured by bioelectrical analysis in infants. Ann Nutr Metab. 2004;48(2):84-9. doi: 10.1159/000077042. Epub 2004 Feb 25. PMID 14988637
- [Background] Galan-Lopez P, Sanchez-Oliver AJ, Pihu M, Gisladottir T, Dominguez R, Ries F. Association between Adherence to the Mediterranean Diet and Physical Fitness with Body Composition Parameters in 1717 European Adolescents: The AdolesHealth Study. Nutrients. 2019 Dec 27;12(1):77. doi: 10.3390/nu12010077. PMID 31892139
- [Background] Henry CJ. Basal metabolic rate studies in humans: measurement and development of new equations. Public Health Nutr. 2005 Oct;8(7A):1133-52. doi: 10.1079/phn2005801. PMID 16277825
- [Background] Garcia-Hermoso A, Vegas-Heredia ED, Fernandez-Vergara O, Ceballos-Ceballos R, Andrade-Schnettler R, Arellano-Ruiz P, Ramirez-Velez R. Independent and combined effects of handgrip strength and adherence to a Mediterranean diet on blood pressure in Chilean children. Nutrition. 2019 Apr;60:170-174. doi: 10.1016/j.nut.2018.08.019. Epub 2018 Oct 18. PMID 30611079
- [Background] Iglesias-Soler E, Rua-Alonso M, Rial-Vazquez J, Lete-Lasa JR, Clavel I, Giraldez-Garcia MA, Rico-Diaz J, Corral MR, Carballeira-Fernandez E, Dopico-Calvo X. Percentiles and Principal Component Analysis of Physical Fitness From a Big Sample of Children and Adolescents Aged 6-18 Years: The DAFIS Project. Front Psychol. 2021 Feb 19;12:627834. doi: 10.3389/fpsyg.2021.627834. eCollection 2021. PMID 33679548
- [Background] WHO Multicentre Growth Reference Study Group. WHO Child Growth Standards based on length/height, weight and age. Acta Paediatr Suppl. 2006 Apr;450:76-85. doi: 10.1111/j.1651-2227.2006.tb02378.x. PMID 16817681
- [Background] Fuentes-Servin J, Avila-Nava A, Gonzalez-Salazar LE, Perez-Gonzalez OA, Servin-Rodas MDC, Serralde-Zuniga AE, Medina-Vera I, Guevara-Cruz M. Resting Energy Expenditure Prediction Equations in the Pediatric Population: A Systematic Review. Front Pediatr. 2021 Dec 6;9:795364. doi: 10.3389/fped.2021.795364. eCollection 2021. PMID 34938700
- [Result] Al-Biltagi M, El Amrousy D, El Ashry H, Maher S, Mohammed MA, Hasan S. Effects of adherence to the Mediterranean diet in children and adolescents with irritable bowel syndrome. World J Clin Pediatr. 2022 Jul 9;11(4):330-340. doi: 10.5409/wjcp.v11.i4.330. eCollection 2022 Jul 9. PMID 36052114